CLINICAL TRIAL: NCT06758453
Title: Bile Acids As Determinants of Postprandial Metabolism
Acronym: PRIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Ministry of Education, Brazil (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jarlei Fiamoncini, Professor PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 73219523.1.0000.0067
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Health; Bile Acid Synthesis Disorders; Postprandial Metabolism; Postprandial Lipids Metabolism
Keywords: Metabolism; Bile Acid; Metabolomics

STUDY DESIGN:
Intervention Model Description: The project aims to map the variability in the appearance of bile acids (BAs) in systemic circulation and explore their role in regulating inflammation and metabolism after meal ingestion. To achieve this, postprandial changes in plasma BA concentrations will be measured in 100 healthy women using a simplified dietary challenge. Capillary blood samples (500 µL) will be collected at 7 time points over 5 hours following the consumption of a high-fat and high-glycemic meal. In the second phase, participants with the highest (n=20) and lowest (n=20) postprandial increases in circulating BAs will be invited for another dietary challenge with the same test meal. During this phase, venous blood samples will be collected to analyze clinical biochemistry markers, the plasma metabolome, signaling molecules (hormones and inflam
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General Population (First Phase) (Experimental): 150 healthy women will participate in the initial assessment of postprandial variability in bile acid (BA) levels after ingesting a test meal.
  Interventions: Other: Dietary Challenge
- High Responders (Second Phase) (Experimental): A subgroup of 20 women with the highest postprandial increase in BA levels from the first phase will undergo further evaluation.
  A subgroup of 20 women with the lowest postprandial increase in BA levels from the first phase will undergo further evaluation.
  Interventions: Other: Dietary Challenge

INTERVENTIONS:
Other: Dietary Challenge — Ingestion of a high-fat, high-glucose meal to induce postprandial variations in bile acids and other metabolic markers.

SUMMARY:
This study aims to understand how bile acids (BAs) appear in the bloodstream after eating and how this might affect inflammation and metabolism. To do this, we will measure changes in BA levels in 100 healthy women after they eat a high-fat and high-carbohydrate meal. Blood samples (a small amount of 500 µL) will be collected from a finger prick at 7 time points over 5 hours. In the second part of the study, 40 women will be invited back-20 with the highest and 20 with the lowest increases in BAs. These participants will eat the same test meal, and blood samples will be taken from a vein to study markers of health, metabolism, inflammation, and the gut microbiome. By exploring how BAs work in the body, this study hopes to find new ways to understand and prevent chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 70 years
* Body mass index (BMI) between 18.5 and 34.9 kg/m²

Exclusion Criteria:

* Pregnant women
* History of bariatric surgery and/or intestinal resection
* Inflammatory bowel disease
* Celiac disease
* Liver disease
* Type 2 diabetes mellitus
* Casein allergy
* Alcohol consumption >30 g/day
* Use of antimicrobial therapy within the past two months

Note: The use of dietary supplements was not considered an exclusion factor. The use of medication for the treatment of chronic diseases was evaluated on a case-by-case basis and did not constitute, a priori, an exclusion factor.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender woman
Enrollment: 150 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma markers of intermediate metabolism and inflammation | 1 day
  Capillary blood samples (approximately 200 µL) were collected after a 12-hour fasting period and at different time points within a 5-hour interval after food intake to assess plasma metabolic and inflammatory markers, such as cytokines (IL-6 and TNF-α [pg/mL]), glucose levels [mg/dL], lipid profile parameters, including triglycerides, total cholesterol, and fractions [mg/dL], as well as bile acids [µmol/L]. These measurements aim to identify the physiological and metabolic responses to food intake.
Cytokines | 1 day
  IL-6 and TNF-α [pg/mL]
Glucose levels | 1 day
  glucose levels [mg/dL]
Lipid profile parameters | 1 day
  triglycerides, total cholesterol, and fractions [mg/dL].
Bile Acids | 1 day
  bile acids [µmol/L]

SECONDARY OUTCOMES:
Urine metabolome | 1 day
  Urine samples were collected after a 12-hours fasting and during the postprandial period (all urine produced during the first 5 hours following food intake) to assess changes in urinary metabolome induced by the intake of the tested meal
24-hour dietary | 1 day
  To assess the participants' food consumption on the day before collection, we applied a 24-hour food recall in which the participant reported everything that was consumed.
Food Frequency Questionnaire (FFQ) | 1 day
  To assess the participants' eating patterns, we applied the quantitative Food Frequency Questionnaire (FFQ) that assesses the participant's food consumption over the last year.
Visual Analog Score (VAS) | 1 day
  The feeling of hunger and satiety will be assessed on a scale of 1 to 10 (arbitrary unit) every hour of the dietary challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No